CLINICAL TRIAL: NCT00828828
Title: Controlled Trial of Serologic Efficacy of Influenza Vaccine in Patients With Sarcoidosis
Brief Title: Antibody Response to Influenza Vaccine in Patients With Sarcoidosis
Acronym: IVS
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Maryam Keshtkar-Jahromi, Clinical Research & DevelopmentCenter, Shaheed Modarres Hospital, Shaheed Beheshti Medical University, Tehran, Iran.
Other Study IDs: SBMU 87-01-120-6003
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Influenza Vaccine; Sarcoidosis; Antibody
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Influenza, Human; Sarcoidosis | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sarcoidosis: Sarcoidosis patients who are assigned to receive influenza vaccine
  Interventions: Biological: Influenza Vaccine
- Healthy Controls: Healthy controls who are assigned to receive influenza vaccine
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — One 0.5 ml dose of influenza vaccine injected intramuscular.
  Other Names: 2008-2009 vaccination campaign of influenza (Solvay Pharma)

SUMMARY:
The purpose of this study is to determine the efficacy of influenza vaccine (antibody response) in patients with sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disease with unclear etiology characterized by the presence of noncaseating granuloma[1]. T helper cells response is exaggerated at the site of disease and cellular immunity depressed in peripheral blood[2]. Cutaneous anergy, lymphopenia and inversion of CD4/CD8 ratio in peripheral blood suggest T helper cells involvement[3].

The action of humeral immune system in sarcoidosis is a matter of controversy. Standard hepatitis B virus vaccination did not provoke protective antibody titer in patients with sarcoidosis[3]. Although antibody response against influenza vaccine in patients with sarcoidosis is not well described, this vaccine is highly recommended in patients with chronic pulmonary diseases such as asthma, COPD and fibrosis [4, 5, 6]. In this study we aim to evaluate the humeral response to the influenza vaccine in sarcoidosis patients and assess vaccine safety.

ELIGIBILITY:
Inclusion Criteria:

Sarcoidosis patients:

* Patients with relevant clinical, radiologic and histologic features of sarcoidosis (all stages).
* Signed informed consent.

Exclusion Criteria:

* Organ failure (kidney, heart, liver).
* Collagen vascular diseases.
* Diabetes.
* Contraindications of vaccine (Egg allergy).
* Patients who receive high dose (> 60 mg/day) steroid therapy.
* Any acute disease.
* Conditions accompanied by immunosuppression (like organ transplantation, HIV).
* Any psychological disease that interferes with regular follow-up.
* Inoculation with influenza vaccine within the past 5 years.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Caes are defined as patients known as sarcoidosis and are under follow up at a tertiary care hospital clinic. Age and sex matched healthy healthcare workers serve as controls.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Serologic Response (equal or more than 4 fold HI titer rise) to each of the 3 antigens of the trivalent vaccine of the 2008-9 influenza vaccine | 4-6 weeks

SECONDARY OUTCOMES:
Magnitude of change in the antibody titer against each of the 3 antigenes of the trivalent vaccine of the 2008/2009 season [A/Brisbane/59/2007(HIN1)-like virus;A/Brisbane/10/2007(H3N2)-like virus;B/Florida/4/2006-like virus] | 4-6 weeks
Protective Antibody (equal or more than 1:40) titer after vaccination | 4-6 weeks
Vaccine Safety (any major or minor side effects) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Keshtkar-Jahromi, MD, MPH, Study Chair — Clinical Research & Development Center, Shahid Modarres Hospital, Shahid Beheshti University (MC), Tehran, Iran; Sasan Tavana, MD, Study Chair — Clinical Research & Developement Center, Shahid Modares Hospital,Shahid Beheshti University (MC), Tehran, Iran; Marzieh Keshtkar-Jahromi, MD, Principal Investigator — Clinical Research & Developement Center, Shahid Modares Hospital, Shahid Beheshti University (MC), Tehran, Iran; Amirsoheil Talebian, MD, Principal Investigator — Clinical Research & Developement Center, Shahid Modares Hospital,Shahid Beheshti University (MC), Tehran, Iran; Mohammad Rahnavardi, MD, Principal Investigator — Clinical Research & Developement Center, Shahid Modares Hospital,Shahid Beheshti University (MC), Tehran, Iran; Talat Mokhtari-Azad, PhD, Principal Investigator — School of Public Health, Tehran University of Medical Sciences, Tehran, Iran
Locations (1):
- Shahid Modarres Hospital, Tehran, Iran

REFERENCES:
- [Background] Newman LS, Rose CS, Maier LA. Sarcoidosis. N Engl J Med. 1997 Apr 24;336(17):1224-34. doi: 10.1056/NEJM199704243361706. No abstract available. PMID 9110911
- [Background] Muller-Quernheim J. Sarcoidosis: immunopathogenetic concepts and their clinical application. Eur Respir J. 1998 Sep;12(3):716-38. doi: 10.1183/09031936.98.12030716. PMID 9762805
- [Background] Mert A, Bilir M, Ozaras R, Tabak F, Karayel T, Senturk H. Results of hepatitis B vaccination in sarcoidosis. Respiration. 2000;67(5):543-5. doi: 10.1159/000067471. PMID 11070460
- [Background] Kmiecik T, Arnoux S, Kobryn A, Gorski P. Influenza vaccination in adults with asthma: safety of an inactivated trivalent influenza vaccine. J Asthma. 2007 Dec;44(10):817-22. doi: 10.1080/02770900701539723. PMID 18097856
- [Background] Ayabe E, Kaneko N, Ohkuni Y, Misawa M, Inoue K, Tanabe Y, Yasui D, Sato C, Mitsuishi Y, Nakashita T, Motojima S. [The efficacy of influenza vaccine for acute exacerbation of chronic obstructive lung disease in elderly patients]. Nihon Kokyuki Gakkai Zasshi. 2008 Jul;46(7):511-5. Japanese. PMID 18700566
- [Background] Wat D, Gelder C, Hibbitts S, Bowler I, Pierrepoint M, Evans R, Doull I. Is there a role for influenza vaccination in cystic fibrosis? J Cyst Fibros. 2008 Jan;7(1):85-8. doi: 10.1016/j.jcf.2007.05.002. Epub 2007 Jul 5. PMID 17616444